CLINICAL TRIAL: NCT01589835
Title: Preventing Diabetes With Facilitated Lifestyle Intervention Prescriptions.Phase 2: Pilot Study
Brief Title: Preventing Diabetes in Those at Risk by Having a Facilitator and Family Doctor Encourage Healthy Activity and Eating Habits
Acronym: FLIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: H12-01330
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Green prescription with facilitator support
  Interventions: Behavioral: Lifestyle changes
- Usual care (Other)
  Interventions: Behavioral: Lifestyle changes

INTERVENTIONS:
Behavioral: Lifestyle changes — Green prescription with support from facilitator

SUMMARY:
Nearly six million Canadians are living with an increased risk of diabetes (prediabetes) and approximately 50% of these will develop type 2 diabetes within five years. The investigators wish to help these people change their lifestyle, to prevent them from getting diabetes. Trials have shown that by supporting people with prediabetes to be more active and have healthier eating habits they can halve their risk. However, these interventions were very costly and not performed in Canada. With the help of local Family Physicians and other health professionals (e.g. physiotherapy, psychology, endocrinology, nursing) the investigators have created a less expensive intervention suitable for the Canadian population and health system. The investigators need to perform a study to see whether these modified approaches are practical for Canadians and likely to be effective. People at risk will be invited to participate from family practices that have helped us in the initial stages of this program. Family practices will be randomized to giving either the study intervention or continue with the physician's usual care. People receiving the intervention will have an appointment with their family doctor to discuss their exercise and eating habits and agree changes that are necessary. A prescription detailing these changes will be completed and signed by the family physician and participant. Participants will be given the name of a lifestyle change facilitator (LCF) who will receive a copy of the prescription and contact the participant to help them set achievable goals. The LCF will contact participants once a month for six months to help them achieve these goals. The investigators eventual aim is to test this intervention in a large-scale randomized control trial. To achieve this it is necessary to pilot all aspects of the trial. Information from the pilot study can then be used to design and perform a large-scale study effectively. The investigators hope that eventually the numbers of Canadians progressing to having diabetes will be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years
* HbA1c of 5.7 to 6.4% and/or FPG of 6.1 to 6.9 mmol/l and/or a 2hr 75g OGTT of between 7.8 and 11.0 mmol/l

Exclusion Criteria:

* People with Type I or II diabetes
* Unstable angina
* Uncontrolled congestive heart failure
* Unstable arrhythmia
* Heart valvular disease
* Severe hypertension (systolic ≥ 200 or diastolic ≥ 120)
* Pregnant women or planning pregnancy within two years
* Life expectancy < 1 year
* Waiting for major surgery
* High risk of fracture
* Pregnancy or planning pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
HbA1c Progression to diabetes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dawes, Principal Investigator — UBC
Locations (1):
- UBC Family Practice, Vancouver, British Columbia, Canada